CLINICAL TRIAL: NCT03358810
Title: Pharyngeal Electrical Stimulation Evaluation for Dysphagia After Stroke
Acronym: PhEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phagenesis Ltd. (Industry)
Collaborators: Regulatory and Clinical Research Institute Inc (Other); Cytel Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHE-05
Record Dates: First submitted 2017-11-21; First posted 2017-12-02 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Dysphagia Following Cerebral Infarction

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active group (Active Comparator): patients randomized to receive active PES
  Interventions: Device: PES
- Sham treatmment (Sham Comparator): Patients randomized to sham will not receive any PES.
  Interventions: Device: PES

INTERVENTIONS:
Device: PES — The PES system is a two-part neurostimulation system. It is composed of a durable component called the Base Station and the single-use sterile disposable Phagenyx® Catheter. The Base Station acts as the user interface and provides the means to generate, optimize and monitor the delivery of electrical stimulation.
  Other Names: Pharyngeal Electrical Stimulation

SUMMARY:
This is a randomized, sham-controlled, patient masked, outcome assessor-blinded study to assess a Pharyngeal Electrical Stimulation (PES) Catheter for treatment of oropharyngeal dysphagia following a stroke.

DETAILED DESCRIPTION:
Randomization will be stratified at each site in a 1:1 fashion. All patients will have the Phagenyx® Catheter placed prior to randomization, and will receive either an active treatment of Pharyngeal Electrical Stimulation (PES) or a sham treatment performed by a health care professional (HCP) that is un-blinded to treatment assignment. All other speech pathology standard dysphagia care will be provided by a speech language pathologist (SLP) that is blinded to treatment assignment. Administration of all protocol-specific assessments will be conducted by personnel blinded to treatment assignment.

The study will follow an adaptive group sequential design with unblinded sample size re-assessment. To ensure 180 evaluable patients with 7-day data and assuming a 20% dropout rate, 225 patients will be enrolled initially. An interim analysis for futility will occur after the first 60 patients complete their 7-day visits and another interim analysis will be performed for efficacy and futility after 120 patients complete their 7-day visits. The total sample size may be increased up to 338 patients after the second interim analysis to ensure up to 270 evaluable patients. Up to 15 investigational centers across the US and possibly Europe will participate in this study. The enrollment period is expected to be approximately 24 months and patient participation will last for approximately 11 weeks. Patients will be assessed at the following intervals: baseline, 48 hours, 7 days, 14 days or at discharge, whichever is first, and 11 weeks after completion of the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 90 years.
* Acute ischemic or hemorrhagic cerebral stroke within 7-28 days of baseline VFSS.
* Score of 0 or 1 on NIHSS question 1a, Level of Consciousness.
* Moderate to severe dysphagia (PAS >4) on baseline VFSS (Baseline VFSS must meet the threshold criteria of demonstrating a PAS of ≥ 4, in three of the six boli (5 mL/1 tsp/bolus), during swallowing "thin liquid" barium media as assessed by the clinical staff administering the VFSS.).
* Willing and able to have the Phagenyx® Catheter placed transnasally.
* Willing and able to provide informed consent.
* Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

* Brainstem stroke.
* Evidence of traumatic brain injury or subarachnoid hemorrhage.
* Other known brain abnormalities documented by history and/or imaging (e.g., tumor, abnormal white matter, inflammatory neuropathy, myelin delamination, hydrocephalus).
* Dysphagia from conditions other than stroke.
* Pre-stroke history of swallowing complaints or treatment or history of diseases known to be associated with swallowing problems (other neurological, head and neck cancer.
* Distorted oropharyngeal anatomy (e.g., pharyngeal pouch, major pharyngeal surgery or head /neck surgery)
* Currently being treatment for pneumonia.
* Mute, global aphasia; no usable speech or auditory comprehension (scores 3 on NIHSS question 9, Best Language)
* NIHSS score of >25
* Presence of a tracheostomy
* Any active implanted device (e.g., cochlear implant, ICD)
* Any progressive neurological disorder (e.g., Parkinson's Disease, Multiple Sclerosis)
* Cognitive impairment that prevents compliance with protocol-specific instructions and assessments
* Unstable cardiopulmonary condition, i.e., not on maintenance therapy.
* Currently participating in another investigational study
* Pregnant or planning to become pregnant while participating in the clinical study -Known Allergy to oral radiographic contrast media (specifically barium) -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-31 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of treatment in reducing the severity of unsafe swallows based on PAS(Penetration Aspiration Scale)of each swallow during VFSS | 48 hours post final treatment
  VFSS (Vidoeflouroscopic Swallow Study) Swallowing safety of a bolus of thin and nectar consistency determined by a videofluoroscopic swallowing study.The PAS provides a scoring mechanism for airway closure and clearance during the VFSS. The PAS is a validated 8-point scale that measures penetration and aspiration. Scores are determined primarily by the depth to which material passes into the airway.
  1. Material does not enter airway
  2. Material enters the airway, remains above the vocal folds, and is ejected
  3. Material remains above the vocal folds, and is not ejected from airway
  4. Material contacts the vocal folds, and is ejected
  5. Material contacts the vocal folds, and is not ejected
  6. Material passes below the vocal folds , and is ejected out airway
  7. Material passes below the vocal folds, and is not ejected from trachea
  8. Material enters the airway , and no effort is made to eject it

SECONDARY OUTCOMES:
To evaluate the efficacy of Phagenyx® treatment in improving nutritional management | 11 weeks post final treatment
  Nutritional management changes will be evaluated via:
  Time from baseline to removal of enteral feeding (i.e., removal of NG tube or PEG or transition to oral feeding, or first diet upgrade,Functional Oral Intake Scale (FOIS) at 7 days, 14 days or discharge, whichever is first, and 11 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Marianjoy, Wheaton, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/10/NCT03358810/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT03358810/SAP_001.pdf